CLINICAL TRIAL: NCT02906501
Title: Effect of Risperidone on Cognitive Functions in Adolescents With ADHD and Behavioral
Brief Title: Effect of Risperidone on Cognitive Functions in Adolescents With ADHD and Behavioral Disturbances
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Ziv Carmel, Principal Investigator, Shalvata Mental Health Center
Other Study IDs: SHA-000-7-16
Record Dates: First submitted 2016-09-11; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: ADHD
Keywords: Risperidone; ADHD; DBD; IGT; CNP; Executive functions
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group I (n=15): Male children and adolescents diagnosed with ADHD not treated with risperidone or any other antipsychotic treatment.
  Interventions: Procedure: The Penn Web-Based Computerized Neurocognitive Battery; Procedure: The Iowa Gambling Test (IGT)
- Group II (n=15): Male children and adolescents diagnosed with ADHD intended to start risperidone or any other antipsychotic treatment due to behavioral problems.
  Interventions: Procedure: The Penn Web-Based Computerized Neurocognitive Battery; Procedure: The Iowa Gambling Test (IGT)
- Group III (n=15): Male children and adolescents diagnosed with ADHD treated with risperidone or any other antipsychotic treatment due to behavioral problems.
  Interventions: Procedure: The Penn Web-Based Computerized Neurocognitive Battery; Procedure: The Iowa Gambling Test (IGT)

INTERVENTIONS:
Procedure: The Penn Web-Based Computerized Neurocognitive Battery — The Battery (PennCNP) of the Brain Behavior Laboratory at the University of Pennsylvania offers a range of probes of human neuropsychological functioning . It was designed for neuropsychological measurement of major cognitive domains. The WebCNP is administered using clickable icons on desktop or laptop computers, in a fixed order. Administrating the tests in a standard fashion fostering optimal performance without aiding the participant is required. For each domain, accuracy and speed are computed. Full battery completion takes approximately 2 hours. Each test begins with a practice module, to assure understanding of the instructions.
Procedure: The Iowa Gambling Test (IGT) — The essential feature of this task is that it mimics real-life situations in the way it factors uncertainty, reward and punishment. The task involves four decks of cards, named A, B, C and D. The goal is to maximize profit on a loan of play money. Subjects are required to make a series of 100 card selections, but are not told ahead of time how many card selections they are going to be allowed to make. Cards can be selected one at a time, from any deck, and subjects are free to switch from any deck to another, at any time and as often as they wish. The decision to select from one deck or another is largely influenced by schedules of reward and punishment. These schedules are pre-programmed and known to the examiner, but not to the subject (Bechara et al., 1994, 1999a).

SUMMARY:
Introduction: The use of low dose risperidone and other antipsychotic drugs off-label as augmentation treatment for adolescents with Attention Deficit Hyperactivity Disorder (ADHD) and Disruptive Behavioral Disorder (DBD) has become widely common worldwide, usually to help control behavioral difficulties. While some argue that agents that block dopaminergic receptors may have a deleterious cognitive effect, others stress their moderating effects, which possibly improve function in all domains, including cognitive functions. Only a few studies have examined this topic, with inconclusive results.

Aim of study: To measure the effect of risperidone treatment on various cognitive functions in a population of ADHD diagnosed children and adolescents with normal IQ.

Design: The study is an observational prospective open label clinical controlled trial. The investigators will compare the performance in a battery of cognitive tasks using the Penn Web-Based Computerized Neurocognitive Battery (WebCNP) and the IGT, in children and adolescents diagnosed with ADHD, with and without risperidone.

Study population: Children and adolescents diagnosed with ADHD, 8-17 years old, may be eligible for this study. We will recruit subjects who their psychiatrist is considering rispieridone treatment, those who are already treated with risperidone and subjects with only stimulants treatment. All pharmacological treatment is supervised and prescribed to subjects by their personal psychiatrist unrelated to the study.

Significance: Better knowledge of the specific cognitive effects of this form of therapy will help us guide both clinical decisions, and recommended monitoring in daily clinical work.

DETAILED DESCRIPTION:
Study Purpose: To evaluate the effect of atypical antipsychotic augmentation, specifically risperidone on specific cognitive domains in adolescents with ADHD and behavioral disturbances.

Hypotheses:

1. Risperidone will improve performance in tasks assessing attention, verbal memory, visual memory and working memory in adolescents with ADHD and DBDs
2. Risperidone will impair performance in tasks assessing spatial memory and some executive functions in adolescents with ADHD and DBDs.
3. Risperidone, but not other atypical antipsychotic, will improve performance on the IGT.

Study Design

General:

This study is an observational prospective open label clinical controlled trial.

The planned study will compare performance, with and without the effect of risperidone, in various cognitive tasks in children and adolescents diagnosed with ADHD.

Each subject will perform a battery of cognitive tasks using the Penn Web-Based Computerized Neurocognitive Battery (WebCNP) and the Iowa Gambling Test (IGT).

Experimental Procedure

Each potential subject and his parents will be screened on the phone for the study. All enrolled subjects will be instructed to avoid taking any stimulant treatment on the days of assessment sessions. On the day of enrolment, each subject will be evaluated by a standard basic medical interview and physical and neurological examinations for evidence of current neurological and physical disorders. They will also be evaluated by the Development and Well-Being Assessment (DAWBA) for evidence of any psychiatric disorders. Parents will also answer DAWBA questionnaire. Subjects who will qualify for the study and their parents will receive a comprehensive explanation on the study and will sign an informed consent form. Subjects will then complete The Penn Web-Based Computerized Neurocognitive Battery (WebCNP) and the Iowa Gambling Test (IGT). The first session will take approximately 2.5 hours. All subjects will undergo a follow up session approximately a month after the first session. The second session will take approximately 2 hours. Subjects in Groups II will be instructed to start taking their risperidone after the first session and on the day of the follow up session. Subjects on Group III will be instructed to take their risperidone or other atypical antipsychotic treatment on days of the experiment in the night before the session at least 8 hours before the sessions and in the month between them. The treatments with Risperidone will be given only according to the decision and guidance of the subject's physician. All subjects will be invited to perform the Penn Continuous Performance Test for a third time, under the influence of their stimulant treatment. Normal IQ will be ascertained using the Raven's Progressive Matrices task which is a part of the WebCNP battery.

ELIGIBILITY:
Inclusion Criteria:

* Male children and adolescents diagnosed with ADHD Age: 8-17 years.
* Psychiatric comorbidities including: Major Depressive disorder, General Anxiety Disorder, Panic Disorder, Obsessive Compulsive Disorder, Oppositional Defiant Disorder, Conduct Disorder, Disruptive Dysregulation Mood Disorder, Intermittent Explosive Disorder and all phobias.

Exclusion Criteria:

* Any current serious medical or surgical illness.
* History of a major neurological illnesses (including brain injury).
* Psychiatric comorbidities including: All psychotic disorders, Bipolar Disorder and personality disorders.
* History of alcohol or substance abuse.
* Intellectual disability: Total IQ< 70

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents diagnosed with ADHD, 8-17 years old, may be eligible for this study. Informed consent will be obtained from potential subjects' parents, and subjects will provide their own assent, according to the local and national IRB committees.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The Penn Web-Based Computerized Neurocognitive Battery (WebCNP) scores | 1 year

SECONDARY OUTCOMES:
Iowa Gambling Task (IGT) scores | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cognition Research Lab Shalvata Mental Hspital, Hod HaSharon, Israel

IPD SHARING:
Plan to Share IPD: Undecided